CLINICAL TRIAL: NCT04896749
Title: Role of Nerve Mobilizations in Decreasing Pain and Disability Among Patients With Cervical Radiculopathy: A Randomized Controlled Trial
Brief Title: Role of Nerve Mobilizations in Decreasing Pain and Disability Among Patients With Cervical Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Momna Asghar, Principal Investigator, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/719-VI/2020
Record Dates: First submitted 2021-04-08; First posted 2021-05-21 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Cervical Radiculopathy
Keywords: cervical radiculopathy; neuromobilization; pain; disability
MeSH Terms: conditions — Radiculopathy; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A/ Nerve mobilization group (Experimental): In this group, patients will receive nerve mobilization exercises along with routine physical therapy. Patients will also be given home plan for cervical isometric exercises.
  Interventions: Other: Nerve mobilization
- Group B/ Conventional physical therapy group (Active Comparator): In this group, patients will receive routine physical therapy and also given home plan for cervical isometric exercises
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Nerve mobilization — Moist pack all over cervical spine for 10 minutes. TENS for 10 minutes at frequency of 60 Hz with 2 electrodes. Cervical traction for 10 minutes with 7 sec hold and 5 sec rest time. Cervical isometric exercises with 7 sec hold and 30 repetitions in each direction twice a day.
  Median, ulnar and radial nerve stretch with 3 sets of 10 repetitions , with 3 sec hold at final stretched position.
  Following nerve mobilizations are used in experimental group/group A:
  Median Nerve: Glenohumeral abduction, wrist extension, supination, glenohumeral lateral rotation, elbow extension, neck lateral bending to opposite side. Radial Nerve: Glenohumeral depression, elbow extension, whole arm internal rotation, wrist flexion Ulnar Nerve: Wrist extension, forearm pronation elbow flexion, glenohumeral lateral rotation, glenohumeral depression, shoulder abduction each with 3 sets of 10 repetitions , with 3 sec hold at final stretched position.
  Arms: Group A/ Nerve mobilization group
Other: Conventional physical therapy — Moist pack for 10 minutes. TENS for 10 minutes at frequency of 60 Hz with 2 electrodes. Cervical traction for 10 minutes with 7 sec hold and 5 sec rest time. Cervical isometric exercises with 7 sec hold and 30 repetitions in each direction twice a day.
  Other Names: Routine physical therapy
  Arms: Group B/ Conventional physical therapy group

SUMMARY:
Objective of the study is to find out the effectiveness of nerve mobilization in patients with cervical radiculopathy. It is a single blinded randomized controlled trial using non-probability convenient sampling. Data is collected from University Physical therapy and Rehabilitation Clinic, University of Lahore, Pakistan.

Alternate hypothesis: There is a significant role of nerve mobilizations in decreasing pain and disability among patients with cervical radiculopathy.

Null hypothesis: There is no significant role of nerve mobilizations in decreasing pain and disability among patients with cervical radiculopathy.

.

DETAILED DESCRIPTION:
It will be a prospectively registered, parallel designed, randomized controlled trial with concealed allocation, conducted in University Physical Therapy and Rehabilitation Clinic, Lahore, Pakistan. Patients who met the eligibility criteria will be informed about the aim of the study. All eligible participants who will agree to participate in the study signed the consent form. Eligibility of the participants will be determined by the two members of the research team before the randomization. After baseline assessment, eligible patients will be randomly assigned (in a 1:1 ratio) into two groups (Group A and Group B). Randomization will be done by one of the research team members using fish bowl method. Randomization assignments will be kept in opaque, sealed envelopes and unsealed by the researchers after baseline testing. Outcome assessor will be masked to group allocation and patients will be instructed not to talk about the content of their exercise program during the post intervention visit and could contact their therapists in case of any problems during trial participation. Help of female physiotherapist will be taken for the female patients. The sample size was calculated as 76 participants (38 per group), allowing statistical power of 80%, an alpha level of 5% and attrition rate of 20% having mean difference of 1.1 and SD of 1.48 and 1.63.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with age between 20 to 45 years
* Patients having pain for more than 4 months
* Patients having positive upper limb neurodynamic test
* Patient with positive spurling test.

Exclusion Criteria:

* Patients with trauma of upper limb and cervical spine
* Dizziness
* Upper limb circulatory disturbance
* Malignancy
* Patients with bilateral symptoms

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Upper extremity functional index (assessing change in ability to do activities with upper limb at baseline and at 4th week of treatment) | Baseline and at 4th week
  It is a patient reported outcome measure used to assess the functional impairment in individuals with upper limb dysfunction. Total score is 80. Greater the score, better the condition of patients.
Numeric pain rating scale (to assess change in pain at between baseline and at 4th week of treatment) | Baseline and at 4th week
  Used for scoring pain level of individual. it is scored 0 to ten.Zero being the lowest pain level, 10 being worst pain level.The patient is asked to make three pain ratings, corresponding to the pain experienced over the past 24 hours.
  The average of the 3 ratings was used to represent the patient's level of pain over the previous 24 hours.
Neck Disability Index scale (to assess the change in disability due to neck pain at baseline and at 4th week of treatment) | Baseline and at 4th week
  This scale is used for accessing how the neck pain is affecting the ability to manage everyday life activities.The NDI can be scored as a raw score or doubled and expressed as a percent. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'. Points of total 10 questions are summed to a total score.Greater score indicates greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Momna Asghar, MSPTN, Principal Investigator — University of Lahore; Muhammad Haider Ullah Khan, MSPTN, Study Chair — University of Lahore
Locations (1):
- University Physical Therapy and Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Information will be shared if needed for betterment and further clinical studies, however the patient's name and personal information will be kept hidden
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after the publication of the study for at least two years
Access Criteria: Data can be accessed by emailing the principal investigator